CLINICAL TRIAL: NCT05829564
Title: Comparison of the Effects of Virtual Reality and Cervical Mobilization in Individuals With Chronic Neck Pain
Brief Title: Virtual Reality and Cervical Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Assist, Prof, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRMOB
Record Dates: First submitted 2023-03-08; First posted 2023-04-25 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain; Virtual Reality
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality+Exercise (Experimental): An exercise program consisting of stretching exercises, posture exercises and breathing exercises and lasting approximately 20-30 minutes will be applied to the individuals in all 3 groups.
  The virtual reality group will performe virtual reality for an additional 20 minutes. (Oculus GO)
  Interventions: Other: virtual reality; Other: exercise
- cervical mobilization+Exercise (Experimental): An exercise program consisting of stretching exercises, posture exercises and breathing exercises and lasting approximately 20-30 minutes will be applied to the individuals in all 3 groups.
  Mobilization techniques that will mobilize the cervical region will be applied to the cervical mobilization group for 20 minutes.
  Interventions: Other: cervical mobilization; Other: exercise
- Control (Other): Control group will only perform an exercise program.
  Interventions: Other: exercise

INTERVENTIONS:
Other: virtual reality — The individuals participating in the study will experience virtual reality.
  Arms: virtual reality+Exercise
Other: cervical mobilization — The individuals participating in the study will be applied cervical mobilization techniques.
  Arms: cervical mobilization+Exercise
Other: exercise — The individuals participating in the study will performed neck-specific exercises.

SUMMARY:
The aim of this study is to compare the effects of virtual reality and cervical mobilization on proprioception, balance parameters, pain, disability level, quality of life and overall felt effect in individuals with chronic neck pain. In addition, it is aimed to qualitatively evaluate the virtual reality perspectives of individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain persisting for at least 3 months
* Being between the ages of 18-65,
* Being sedentary (not included in any physical therapy program in the last 6 months), ->10 points from the Neck Disability Index

Exclusion Criteria:

* History of previous spinal surgery
* Neurological, cardiopulmonary, musculoskeletal disease affecting physical performance
* Any pathology in the shoulder joint
* Spinal trauma history
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Joint position sense error | Change from Baseline balance after 4 weeks/10 sessions.
  Proprioception in all cervical directions will assessed by Cervical Range of Motion device.
Baropodometer assessments-Pressure distribution | Change from Baseline proprioception after 4 weeks/10 sessions.
  Pressure distribution will assess with FreeMed baropodometric platform and will record as percentage.
Baropodometer assessments- Center of gravity | Change from Baseline proprioception after 4 weeks/10 sessions.
  Center of gravity will assess with FreeMed baropodometric platform and will record as mm.
Baropodometer assessments- Oscillations | Change from Baseline proprioception after 4 weeks/10 sessions.
  Oscillations will assess with FreeMed baropodometric platform.
Baropodometer assessments- Sway velocity | Change from Baseline proprioception after 4 weeks/10 sessions.
  Sway velocity will assess with FreeMed baropodometric platform and will record as degrees.
Functional Balance | Change from Baseline proprioception after 4 weeks/10 sessions.
  10 meter walking speed and four square step-test will be combined to report dynamic balance.

SECONDARY OUTCOMES:
Cervical Pain | Change from Baseline cervical pain after 4 weeks/ 10 sessions.
  Visual Analog Scale will be used to assess this outcome measure.
Functional disability | Change from Baseline functional disability after 4 weeks/ 10 sessions.
  Neck Disability Index will be used to assess this outcome measure.
quality of life about cervical pain | Change from Baseline quality of life about cervical pain after 4 weeks/ 10 sessions.
  SF-36 will be used to assess this outcome measure.
Global perceived effect | Change from Baseline Global perceived effect after 4 weeks/ 10 sessions.
  Global perceived effect scale will be used to assess this outcome measure/ 10 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Oge, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No